CLINICAL TRIAL: NCT03762447
Title: A Phase 1 Study Exploring the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INCB086550 in Participants With Advanced Solid Tumors
Brief Title: A Study Exploring the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INCB086550 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 86550-102; 2019-004377-27 (EudraCT Number)
Record Dates: First submitted 2018-11-19; First posted 2018-12-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
Keywords: solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB086550 (Experimental)
  Interventions: Drug: INCB086550

INTERVENTIONS:
Drug: INCB086550 — INCB086550 will be orally administered once or twice daily in continuous or intermittent dose schedules.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics, and early clinical activity of INCB086550 in participants with advanced solid tumors who have failed prior treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumors with measurable lesions per RECIST v1.1 or RANO for primary brain tumors that are considered nonamenable to surgery or other curative treatments or procedures. Tumor lesions located in a previously irradiated area, or in an area subjected to other loco-regional therapy, are considered measurable per RECIST v1.1 if progression has been demonstrated in the lesion.
* Willingness to undergo a tumor biopsy to obtain tumor tissue,Pretreatment and on-treatment tumor biopsies are required.
* Must have disease progression after treatment with available therapies that are known to confer clinical benefit or who are intolerant to or ineligible for standard treatment. There is no limit to the number of prior treatment regimens.
* Eastern Cooperative Oncology Group performance status score of 0 or 1.
* Life expectancy > 12 weeks.
* Willingness to avoid pregnancy or fathering children.
* Part 2 Expansion Cohort 2-A only: Participants with any type of solid tumor that has a local regulatory approval for an anti-PD-1 therapy. Other tumor types may be enrolled with medical monitor approval. Participants must have had confirmed disease progression on a prior anti-PD-1 monoclonal antibody.
* Part 2 Expansion Cohort 2-B only: Participants with select solid tumors who are immunotherapy-naïve.
* Part 3 MSI-H or dMMR Expansion Cohort only (Enrolled ex-United States only): Participants with any MSI-H or dMMR solid tumor who are immunotherapy-naïve.
* Part 4 HPV-driven expansion cohort only: Participants with any HPV-positive solid tumor who have received prior standard therapy.

Note: HPV-positive status determined by a local laboratory using p16 IHC, polymerase chain reaction methods, or other locally-available method to detect HPV

Exclusion Criteria:

* Laboratory values not within the Protocol-defined range.
* Clinically significant cardiac disease.
* History or presence of an ECG that, in the investigator's opinion, is clinically meaningful.
* Untreated brain or central nervous system (CNS) metastases or brain or CNS metastases that have progressed. Participants who have previously treated and clinically stable brain or CNS metastases and have not required steroids for at least 7 days before study treatment are eligible.
* Known additional malignancy that is progressing or requires active treatment.
* Has not recovered to ≤ Grade 1 or baseline from toxic effects of prior therapy and/or complications from prior surgical intervention before starting study treatment.
* Treatment with anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Active infection requiring systemic therapy.
* Active HBV or HCV infection that requires treatment.
* Known history of HIV (HIV 1/2 antibodies).
* Known hypersensitivity or severe reaction to any component of study drug or formulation components.
* Prior receipt of an anti-PD-L1 therapy for all participants.
* Presence of a gastrointestinal condition that may affect drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Baseline through 90 days after end of treatment, estimated up to 12 months.
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCB086550 in fasted and food effect conditions | Approximately 1 month
  Maximum observed plasma or serum concentration.
tmax of INCB086550 in fasted and food effect conditions | Approximately 1 month
  Time to maximum concentration.
AUC0-tau of INCB086550 in fasted and food effect conditions | Approximately 1 month
  Area under the plasma or serum concentration-time curve from time = 0 to the end of dosing period at steady state
AUC 0-t and/or AUC0-∞ of INCB086550 in fasted and food effect conditions | Approximately 1 month
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration, or Area under the single-dose plasma concentration-time curve from Hour 0 to infinity
t½ of INCB086550 | Approximately 1 month
  Apparent terminal-phase disposition half-life.
λz of INCB086550 | Approximately 1 month
  Apparent terminal-phase disposition rate constant
CL/F of INCB086550 | Approximately 1 month
  Apparent oral dose clearance.
Vz/F of INCB086550 | Approximately 1 month
  Apparent oral dose volume of distribution.
Pharmacokinetic/pharmacodynamics correlation | Approximately 1 month
  Evaluation of the ability of INCB086550 to modulate PD-L1 expression levels as assessed by flow cytometry protein analyses.
Objective response rate | Every 8 weeks for the duration of study participation; estimated to be 12 months.
  Defined as the percentage of participants having complete response (CR) or partial response (PR) by investigator assessment of radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or response assessment in Neuro-Oncology (RANO).
Disease control rate | Every 8 weeks for the duration of study participation; estimated to be 12 months.
  Defined as the percentage of participants having CR, PR, or stable disease ≥ 12 weeks by investigator assessment of radiographic disease assessments per RECIST v1.1 or response assessment in Neuro-Oncology (RANO).
Duration of response | Every 8 weeks for the duration of study participation; estimated to be 12 months.
  Defined as the time from the first documented evidence of CR or PR until the earliest date of disease progression by investigator assessment per RECIST v1.1 for response assessment in Neuro-Oncology (RANO), or death due to any cause, if occurring sooner than progression.
Cmin of INCB086550 in fasted and food effect conditions | Approximately 1 month
  Minimum observed plasma or serum concentration of INCB086550

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Hayer, MD, PhD, Study Director — Incyte Corporation
Locations (25):
- United States (7):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Tampa, Florida
  - Aamc Oncology and Hematology, Annapolis, Maryland
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- France (4):
  - Chu Hopital de La Timone, Marseille
  - Icm Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut Universitaire Du Cancer de Toulouse Oncopole, Toulouse
- Italy (5):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - European Institute of Oncology, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Napoli
  - Irrcs Instituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria Alle Scotte, Siena
- United Kingdom (5):
  - Addenbrooke'S Hospital, Cambridge
  - Guys and St Thomas Nhs Foundation Trust, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koblish HK, Wu L, Wang LS, Liu PCC, Wynn R, Rios-Doria J, Spitz S, Liu H, Volgina A, Zolotarjova N, Kapilashrami K, Behshad E, Covington M, Yang YO, Li J, Diamond S, Soloviev M, O'Hayer K, Rubin S, Kanellopoulou C, Yang G, Rupar M, DiMatteo D, Lin L, Stevens C, Zhang Y, Thekkat P, Geschwindt R, Marando C, Yeleswaram S, Jackson J, Scherle P, Huber R, Yao W, Hollis G. Characterization of INCB086550: A Potent and Novel Small-Molecule PD-L1 Inhibitor. Cancer Discov. 2022 Jun 2;12(6):1482-1499. doi: 10.1158/2159-8290.CD-21-1156. PMID 35254416